CLINICAL TRIAL: NCT04048343
Title: A 52-Week, Open-Label, Multicentre Study to Evaluate the Safety of Tezepelumab in Japanese Adults and Adolescents With Inadequately Controlled Severe Asthma (NOZOMI)
Brief Title: Long-term Safety of Tezepelumab in Japanese Subjects With Inadequately Controlled Severe Asthma
Acronym: NOZOMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5180C00019
Record Dates: First submitted 2019-06-05; First posted 2019-08-07 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Severe Asthma
Keywords: Asthma; Uncontrolled Asthma; Severe Uncontrolled Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: All subject will be dosed tezepelumab administered subcutaneously
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tezepelumab (Experimental): Tezepelumab: Tezepelumab subcutaneous injection
  Interventions: Drug: Biological: Experimental: Tezepelumab

INTERVENTIONS:
Drug: Biological: Experimental: Tezepelumab — Tezepelumab subcutaneous injection every 4 weeks
  Other Names: Tezepelumab

SUMMARY:
This is an open-label, single arm study designed to evaluate the safety of tezepelumab administered subcutaneously every 4 weeks in Japanese adult and adolescent subjects with inadequately controlled severe asthma.

DETAILED DESCRIPTION:
This is open-label, single arm study designed to evaluate the safety of tezepelumab in adults and adolescents with severe, uncontrolled asthma on medium to high-dose ICS and at least one additional asthma controller medication with or without OCS. Approximately 66 subjects will be dosed in Japan. Subjects will receive tezepelumab administered via subcutaneous injection at the study site, over a 52-week treatment period. The study also includes a post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Age. 12-80 Documented physician-diagnosed asthma for at least 12 months Subjects who have received a physician-prescribed asthma controller medication with medium or high dose ICS for at least 12 months.

Documented treatment with a total daily dose of either medium or high dose ICS (≥ 500 µg fluticasone propionate dry powder formulation equivalent total daily dose) for at least 3 months.

At least one additional maintenance asthma controller medication is required according to standard practice of care and must be documented for at least 3 months.

Documented history of at least 1 asthma exacerbation events within 12 months. ACQ-6 score ≥1.5 at screening or on day of registration.

Exclusion Criteria:

Pulmonary disease other than asthma. History of cancer. History of a clinically significant infection. Current smokers or subjects with smoking history ≥10 pack-yrs. History of chronic alcohol or drug abuse within 12 months. Hepatitis B, C or HIV. Pregnant or breastfeeding. History of anaphylaxis following any biologic therapy. Subject randomized in the current study or previous tezepelumab studies

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaharu Shinkai, MD, Principal Investigator — Tokyo Shinagawa Hospital Medical Corporation Association, Japan
Locations (4):
- Japan (4):
  - Research Site, Chūōku
  - Research Site, Sagamihara-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00019&attachmentIdentifier=97c43e3b-e498-4f8b-85d5-2faf4536e7c7&fileName=D5180c00019_CSP-v3_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00019&attachmentIdentifier=0c96c5d1-f13b-49eb-9068-8e12565da16d&fileName=D5180c00019_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00019&attachmentIdentifier=a5b1e7be-72d8-4ca7-ae06-a71b18e628ec&fileName=D5180c00019_SAP-v3_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 subjects fulfilled all inclusion and exclusion criteria and were registered to receive treatment at 5 centres in Japan.
Pre-assignment Details: All registered subjects received treatment.
Groups:
- Tezepelumab 210mg Q4W: Tezepelumab admistered every 4 weeks subcutaneously
Period: Overall Study
Arm/Group | Tezepelumab 210mg Q4W
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tezepelumab 210mg Q4W
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 52
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 0
  Black or African American | 0
  Asian | 65
  Native Hawaiian or Other Pacific Islander | 0
  American Indian or Alaska Native | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: The number of subjects who experienced an AE during on-treatment period was summarised.
Time Frame: From first dose of study drug until last study visit at Week 64
Measure: Count of Participants; unit: Participants
Groups:
- Tezepelumab 210 Q4W: Tezepelumab administered every 4 weeks subcutaneously
Arm/Group | Tezepelumab 210 Q4W
Number analyzed (Participants) | 65
Participants | 39

ADVERSE EVENTS:
Time Frame: From first dose of study drug until last study visit at Week 64
Arm/Group | Tezepelumab 210mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 4/65
Other Adverse Events (participants affected / at risk) | 29/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab 210mg Q4W (N=65)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab 210mg Q4W (N=65)
Injection site erythema (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 13 (18)
Oral herpes (Infections and infestations) | 2 (4)
Pharyngitis (Infections and infestations) | 6 (6)
Rhinitis (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT04048343/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT04048343/SAP_001.pdf